CLINICAL TRIAL: NCT03120377
Title: Respiratory and Musculoskeletal Effects After a Whole Body Vibration Training Program in Adult Renal Transplant Recipients: A Randomized Controlled Trial
Brief Title: Efficiency of a Whole Body Vibration Training Program in Adult Renal Transplanted Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Lívia Gomes da Rocha, physiotherapist of the post-graduation program in physiotherapy of the Federal University of Pernambuco, principal investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LRocha
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Kidney Transplantation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platform group (Active Comparator): Group submitted to the whole body vibration training program
  Interventions: Other: Platform
- Platform sham group (Sham Comparator): Group that will receive the whole body vibration simulation treatment without the therapeutic effect of the platform, but with vibrating platform connected with the display on and a sound device coupled with vibration-generated noise recording, but without therapeutic purposes.
  Interventions: Other: Platform sham

INTERVENTIONS:
Other: Platform — Whole body vibration training will consist of 12 consecutive weeks with two sessions per week on alternate days. Initially, before training with the vibratory platform, stretches lasting 5 to 10 minutes will be performed, with a series of 60 seconds for each of the following muscle groups: pectorals, sternocleidomastoids, scalenes, quadriceps and ischiatibial muscles. Patients will be monitored through vital signs for follow-up.
  Arms: Platform group
Other: Platform sham — will receive the treatment without the therapeutic effect of the platform, but with vibrating platform connected with the display lit and a sound device coupled with a noise recording generated by the vibration, but without therapeutic purposes.
  Arms: Platform sham group

SUMMARY:
Evaluate the effectiveness of a Whole body vibration training program on quadriceps muscle strength, functional capacity and respiratory muscle strength in adult renal transplant recipients

DETAILED DESCRIPTION:
The study will be a randomized controlled clinical trial involving adult renal transplant recipients, who will be recruited through eligibility criteria at Nephrology outpatient clinics of the Kidney Transplantation Centers of the Hospital das Clínicas of the Federal University of Pernambuco (HC-UFPE). Individuals will be randomized and assigned to one of the following groups: Platform Group, which will perform 12-week whole body vibration training or Platform SHAM Group that will receive treatment without the therapeutic effect of the platform. Afterwards, the patients will be submitted to an evaluation, a form with sociodemographic data, the clinical history of the disease and the laboratory tests will be completed, after which the pulmonary function, respiratory muscle strength, quadriceps muscle strength and thickness, postural balance , Functional capacity, quality of life, risk of falls and level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* patients with more than 1 year of kidney transplant surgery
* stable graft function (creatinine <1.8 mg / dL)
* hemoglobin> 8g / dL
* age range 18 And 59
* both sexes

Exclusion Criteria:

* PAS> 160mmHg and PAD> 100mmHg
* Patients with neurological, diagnosed or pulmonary heart disease
* Involved in some physiotherapeutic program
* With hospitalization history for 3 months
* Pregnant
* Current or previous smokers
* That use pacemaker, screws and / or pins in the body
* Presence of acute migraines, labyrinthitis
* History of thrombosis
* Body weight greater than 120Kg
* Cognitive, visual and / or auditory deficits
* Osteomioarticular diseases that would impair evaluation procedures and / or training

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-10-23 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle strength | 20 minutes
  Will be performed the examination of the Maximum Voluntary Isometric Contraction
Functional capacity | 10 minutes
  The 6-minute walk test will be used
Respiratory muscle strength | 20 minutes
  Will be performed through the manocacuometry with the evaluation of the maximum respiratory pressures

SECONDARY OUTCOMES:
Thickness of the quadriceps | 10 minutes
  This measure will be obtained through the portable Ultrasound
Postural balance | 20 minutes
  The static and dynamic postural balance will be evaluated through the Biodex Balance System
Pulmonary function | 15 minutes
  Slow and forced spirometry will be used
Risk of fall | 5 minutes
  The International Fall Efficiency Scale (FES-I) will be used
Level of physical activity | 5 minutes
  It will be evaluated by the International Physical Activity Questionnaire
Quality of life | 10 minutes
  Will be applied the Medical Outcomes Study Quality of Life Questionnaire - Short-Form Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Lívia Rocha, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Laboratório Cardiopulmonar, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided